CLINICAL TRIAL: NCT04469738
Title: Evaluating a Treatment Effect in Patients With FBSS Using an Electronic Nose: a Pilot Study
Acronym: NOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: the eNose company (Unknown)
Responsible Party: Principal Investigator, Moens Maarten, principal investigator, Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: NOSE
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Failed Back Surgery Syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCS off (Experimental)
  Interventions: Device: SCS is switched off
- SCS on (Experimental)
  Interventions: Device: SCS is switched on

INTERVENTIONS:
Device: SCS is switched off — Spinal cord stimulator is switched off for 12 hours
  Arms: SCS off
Device: SCS is switched on — Spinal cord stimulator is functioning
  Arms: SCS on

SUMMARY:
This study is an experimental single-center pilot study investigating Volatile Organic Compounds patterns in exhaled breath during on and off states of SCS, in patient with Failed Back Surgery Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FBSS (Failed conservative treatments for pain including but not limited to pharmacological therapy and physical therapy) and currently being treated with spinal cord stimulation.

Exclusion Criteria:

* Patients with a diagnosis of cancer.
* Patients with major psychiatric problems.
* Patients with an underlying respiratory disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-03-27 (Actual); Study Completion 2021-03-27 (Actual)

PRIMARY OUTCOMES:
Exhaled breath changes | Two times on the same day; once while SCS is switched off and once while SCS is switched on. Total study duration lasts one day.
  The investigators will examine the difference in exhaled breath patterns between both measurements (SCS on versus SCS off), measured with the Aeonose.

SECONDARY OUTCOMES:
Pain intensity scores using the Visual Analogue Scale | Two times on the same day; once while SCS is switched off and once while SCS is switched on. Total study duration lasts one day.
  Pain intensity score on that time on a Visual Analogue Scale (VAS) ranging from zero (no pain) towards 10 (worst possible pain) for the pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Moens, Prof. dr., Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Belgium